CLINICAL TRIAL: NCT03667833
Title: The Effect of Shoulder Brace on Muscle Activation and Scapular Kinematics in Patients With Shoulder Impingement Syndrome and Rounded Shoulder Posture
Brief Title: Shoulder Brace on Muscle Activation and Scapular Kinematics in Patients With Shoulder Impingement Syndrome and Rounded Shoulder Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201805043RINC
Record Dates: First submitted 2018-08-16; First posted 2018-09-12 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-06

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Shoulder Brace
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shoulder brace with comfortable tension (Experimental): Self-comfortable tension of strap will be adjusted by subject's feedback with comfortable feeling as "please feel postural correction by shoulder brace without tight pressure".
  Interventions: Other: Shoulder brace
- shoulder brace with forced tension (Experimental): Forced tension, the self-comfortable tension of strap will be increased till forced tension of strap using buckles.
  Interventions: Other: Shoulder brace

INTERVENTIONS:
Other: Shoulder brace — Shoulder brace is a designed elastic strap to correct scapula alignment in different characteristics such as tension and direction of force.

SUMMARY:
Background:

Rounded shoulder posture (RSP), associated with altered scapular kinematics and imbalance of muscle activation, is one of potential risks for shoulder impingement syndrome (SIS) due to alignment deviation of scapula. Evidence showed shoulder brace improved degree of RSP by postural correction. However, it is unknown whether shoulder brace with different characteristics (tension and direction) is optimal for muscle activation and scapular kinematics in patients with SIS and RSP.

Objective:

There are 4 objectives for the present study: (1) to investigate the relationships among degree of RSP, scapular kinematics and muscle activation in SIS patients with RSP; (2) to compare the effect of shoulder brace on degree of RSP, muscle balance ratios (Upper trapezius/Lower trapezius, Upper trapezius/ Serratus anterior) and scapular kinematics (upward/downward rotation, anterior/posterior tilt, external/internal rotation) during arm movements; (3) to compare the effect of two tensions of brace strap (self-comfortable and forced tension) in symptomatic impingement patients with RSP; (4) to compare the effect of two types of direction of strap (paraspinal muscle and diagonal orientation) in symptomatic impingement patients with RSP.

Design:

Patients with SIS and RSP will be recruited in this study. Participants will be randomly assigned into 2 groups (self-comfortable following forced tension and forced following self-comfortable tension groups) with 2 directions of strap in each tension wearing shoulder brace. Each patient has the assessment 2 times with 1-week interval. Pectoralis minor, acromial distance, scapular index and shoulder angle will be used to assess degree of RSP. Three-dimensional electromagnetic motion analysis and electromyography muscle activity will be used to record the scapular kinematic, absolute muscle activation and muscular balance ratios during arm movements with or without shoulder brace.

Main outcome measures:

Scapula kinematic (upward/downward rotation, anterior/posterior tilt, external/internal rotation), absolute muscle activation (Upper trapezius, Middle Trapezius, Lower trapezius, Serratus anterior) and muscle balance ratios (Upper trapezius/Lower trapezius, Upper trapezius/Serratus anterior) are main outcomes of the study.

DETAILED DESCRIPTION:
Participants will be recruited from outpatient clinic in National Taiwan University Hospital (NTUH) and also through general announcements in social media. Subjects will be undergoing physical examinations for eligibility by a physical therapist. Thoracic kyphosis angle, one inclinometer over 1st and 2nd thoracic spines, and another inclinometer over the 12th thoracic and 1st lumbar spines in relaxed standing with adopting a natural posture of the subject, is calculated by the summation of the angle recorded by two inclinometers. Participants will sign a consent form approved by the National Taiwan University Hospital institutional review boards. Participant characteristics will be collected by the assessor including age, gender, height, weight, dominant side, involved side, VAS (Visual Analogue Scale) pain intensity during arm movements, symptom duration and shoulder function. Shoulder function will be assessed by Flexilevel Scale of Shoulder Function (FLEX-SF), a self-administered questionnaire. The questionnaire was commonly used in shoulder pain patients to assess shoulder function with sufficient psychometric properties. Lower FLEX-SF score represents limited function.

Subjects will be randomly assigned into 2 groups (self-comfortable following forced tension and forced following self-comfortable tension groups) with 2 directions of strap in each tension wearing shoulder brace. Each subject has the assessment 2 times with 1-week interval. At the first, each subject will be assessed on PMI, SI, AD and SA with and without shoulder brace in resting position. Then the surface EMG electrodes and FASTRAK kinematic sensors will be attached to the subjects. Surface EMG electrodes will be placed on upper trapezius, middle trapezius, lower trapezius and serratus anterior of involved shoulder. Three electromagnetic sensors will be attached to the sternum, the flat bony surface of the acromion and the distal humerus via Velcro straps.

Then subject will be tested wearing shoulder brace with two tensions of strap (self- comfortable/ forced) under two directions of strap (paraspinal muscle/ diagonal orientation). Strap is applied from mid-level of thoracic spinal process to mid-point of clavicle on the tested side and then pulled downward diagonally back to the thoracic spinal process and then applied the same way in the other side. In general, strap had a cross on mid-thorax and ran through mid-point of clavicle and axillary two sides. For the strap tension, length of strap will be adjusted with buckles relative to original length of figure 8 by the experimenter. Self- comfortable tension of strap will be adjusted by subject's feedback with comfortable feeling as "please feel postural correction by shoulder brace without tight pressure". Accordingly, the self-comfortable tension of strap will be increased till forced tension of strap using buckles. Direction of strap will change bilaterally as upper part of shoulder brace is fixed at 2 points of shoulder brace .

Then subjects will be tested and familiarized with the arm movement with and without shoulder brace. To ensure that each subject perform arm movements at a standard speed, a metronome will be set as one beat per second. Subjects will be asked to elevate and lower arm by following three beats, respectively. Each subject will do task three times with or without shoulder brace in each session. After one week from the first assessment, each subject will be assessed again under another condition of strap tension according to their assignment groups.

Maximum voluntary isometric contraction (MVIC) of the subject will be collected after the testing session to prevent fatigue of the scapular muscles. The MVIC for upper trapezius muscle will be measured during resisted shoulder flexion. The subjects will be seated with shoulder flexion 90 degrees and resistance will be applied on the distal arm. For measuring MVIC of middle trapezius muscle, the subjects will lie prone with testing arm at 90 degrees of abduction. For measuring MVIC of lower trapezius muscle, the subjects will lie prone with testing arm at 120 degrees of abduction in line with muscle fibers. Resistances will be applied to against further elevation. For measuring MVIC of serratus anterior muscle, the subjects will be seated with arm elevated at 135 degrees. Resistances will be applied to distal upper arm against further elevation. The MVICs will be collected for 5 seconds for 3 trials, with a 1- minute rest interval between each trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 of the following 5 impingement signs

  1. Neer's impingement test;
  2. Hawkins-Kennedy impingement test;
  3. Empty can test;
  4. External resisted test;
  5. Pain during rotator cuff palpation
* Acromial distance higher than 2.6 cm.

Exclusion Criteria:

* History of shoulder dislocation, fracture, shoulder surgery, or direct contact injury to the neck or upper extremities within the past 3 months
* Glenohumeral joint instability (apprehension test or sulcus sign)
* Neurological disorders (thoracic outlet syndrome or pectoralis minor syndrome)
* Pain (VAS>5) during the experimental tasks
* Excessive thoracic kyphosis higher than 50 degrees

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Scapular kinematics | 1 year
  This study will follow the ISB guidelines for constructing a shoulder joint coordinate system. Scapular orientation relative to the thorax will be described using a Euler angle sequence of rotation about Zs (protraction/retraction), rotation about Y's (downward /upward rotation), and rotation about X"s (posterior/anterior tipping).
  Unit of measure is degree.
Surface Electromyography of shoulder muscle | 1 year
  The mean sEMG amplitude of each muscle reported as a percentage of MVIC will be used to describe the activity of upper trapezius, middle trapezius, lower trapezius and serratus anterior muscle.
  Unit of measure is percentage of maximal voluntary isometric contraction.

SECONDARY OUTCOMES:
Pectoralis minor index (PMI) | 1 year
  PMI is used to measure the length of the PM. The subjects will be seated erect with their test arms by side. Forearm position is neutral with hand in resting position. The measurement of PM muscle length is from the medial-inferior angle of the coracoid process to the sternocostal junction of the inferior aspect of the fourth rib with a caliper. The PMI is calculated by dividing he resting muscle length by the subject's height and multiplying by 100.
  Unit of measurement is percentage because length and height have been divided each other.
Acromial distance (AD) | 1 year
  Acromial distance is defined as the distance from table to border of lateral-inferior acromion when subjects are in supine position with shoulder in neutral position (Host HH, 1995). A score≧ 2.6 cm will be defined as RSP.
Scapular index (SI) | 1 year
  SI was determined by measuring the distance from the mid-point of the sternal notch (SN) to the medial aspect of the coracoid process (CP) and the horizontal distance from the posterolateral angle of the acromion (PLA) to the thoracic spine (TS) with a soft tape measure. The subjects will be seated in upright position with their test arms by side (Borstad JD, 2006). The SI is calculated by dividing the SN-CP length by the PLA-TS length and multiplying by 100.
  PMI is used to measure the length of the PM. The subjects will be seated erect with their test arms by side. Forearm position is neutral with hand in resting position. The measurement of PM muscle length is from the medial-inferior angle of the coracoid process to the sternocostal junction of the inferior aspect of the fourth rib with a caliper. The PMI is calculated by dividing he resting muscle length by the subject's height and multiplying by 100.
  Unit of measurement is percentage because length have been divided each other.
Shoulder angle (SA) | 1 year
  The angle formed at the intersection of the line between the midpoint of the humerus and spinous process of C7 and the horizontal line through the midpoint of the acromial process, reflects anterior translation of shoulder in sagittal plane.
Self-reported flexilevel scale of shoulder function (FLEX-SF) | 1 year
  The selection of the FLEX-SF scale to assess shoulder function and disability in this study is based on its entire continuum assessment of shoulder functions and appropriate psychometric properties of reliability, validity, and responsiveness to clinical change. In this scale, respondents answer a single question that grossly classifies their level of function as low, medium, or high. They then respond to only the items that target their level of function. Scores will be recorded from 1, with the most limited function, to 50, without any limited function in the subject.
  Unit of measurement is purely score.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Jenq Lin, Phd, Study Chair — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan